CLINICAL TRIAL: NCT01479907
Title: Synbiotics and Gastrointestinal Function Related Quality of Life After Colectomy for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George Theodoropoulos, Ass Professor of Surgery, Athens Medical School, University of Athens
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SYNBIOTICSCOLON
Record Dates: First submitted 2011-11-16; First posted 2011-11-28 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synbiotics (Active Comparator): A specific multistrain/multifi ber synbiotic composition of prebiotics and probiotics (Synbiotic Forte™, "IONIA" Pharmaceuticals, Athens, Greece) was administered at the active comparator arm of the study. It contained 10 [11] of each of four lactic acid bacteria (LAB): Pediococcus pentosaceus 5-33:3, Leuconostoc mesenteroides 32-77:1, Lactobacillus paracasei ssp. paracasei 19, and Lactobacillus plantarum 2362, and 2.5 g of each of the four fermentable fibers (prebiotics): b-glucan, inulin, pectin and resistant starch. The synbiotics were delivered in sachets and then mixed with water (12 g in 250 mLof water once daily). Th e treatment started on the day patients tolerated per os liquid intake (2nd-4th POD). The intervention period lasted 15 days.
  Interventions: Dietary Supplement: Synbiotics
- Placebo (Placebo Comparator): The patients belonging to the placebo comparator arm received only the 4 fi bers and no LAB (12 gin 250 mLof water once daily for 15 days). All the subjects were interviewed by a dedicated research fellow (KP) and reactions to the product, and any adverse events occurring in the 15-day period were recorded.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotics — 12 gr in 250 cc of water once daily X 15 days
  Arms: Synbiotics
Dietary Supplement: Placebo — 12 gr in 250 cc of water once daily X 15 days
  Arms: Placebo

SUMMARY:
The aim of this double-blinded prospective randomised trial is to explore the potential benefits of early postoperative administration of Synbiotics (combination of prebiotics and probiotics) to patients who have undergone colectomy for cancer. The patients are randomised to either synbiotics or placebo administration at the day they are able to tolerate po liquid diet and for 15 days thereafter.

Primary end points of the study will be:

Assessment of gastrointestinal function-related quality of life at 1, 3 and 6 months postoperatively by the use of the validated questionnaire GIQLI (Gastrointestinal Quality of Life Index)

Secondary end points will be:

-Assessment of functional bowel disorders (diarrhea, constipation, etc) at 1, 3 and 6 months postoperatively based on the respective domains of the validated instrument EORTC QLQ-C30

DETAILED DESCRIPTION:
The study patients are randomized before surgery to receive either synbiotics (Synbiotics group) or placebo (Control group). Equal randomization is accomplished using a computer-generated random allocation schedule. The method of allocation concealment is sequentially numbered sealed opaque envelopes technique. Both synbiotics and placebo preparations are in foil-sealed sachets stored in identical numbered containers. Both study products are white powders, identical in weight, smell, and taste. Thus, the identity of the specific product is blind to participants, support staff and investigators for the entire duration of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Colectomy for histologically proven colorectal adenocarcinoma

Exclusion Criteria:

* Pregnancy,
* hereditary cancer,
* history of inflammatory bowel disease,
* metastatic disease at presentation,
* emergency operation,
* major postoperative complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Assessment of gastrointestinal function-related quality of life at 1, 3 and 6 months postoperatively | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: George E Theodoropoulos, Principal Investigator — University of Athens
Locations (1):
- First Department of Propaedeutic Surgery of Athens Medical School, Hippocration General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No